CLINICAL TRIAL: NCT04941612
Title: Use of the Bioabsorbable Activa IM-Nail™ in Pediatric Diaphyseal Forearm Fractures: a Cohort Study of 30 Patients
Brief Title: Use of the Bioabsorbable Activa IM-Nail™ in Pediatric Diaphyseal Forearm Fractures
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Children's Fractures Interest Group, Denmark (Other)
Responsible Party: Principal Investigator, Morten Jon Andersen, Consultant Orthopedic Surgeon, Children's Fractures Interest Group, Denmark
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H-21004012
Record Dates: First submitted 2021-05-24; First posted 2021-06-28 (Actual); Last update posted 2021-06-28 (Actual); Status verified 2021-06

CONDITIONS: Fracture Fixation, Intramedullary; Forearm Fracture; Fracture Healing; Child, Only; Implant Complication

STUDY DESIGN:
Intervention Model Description: Cohort study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Activa IM-Nail (Experimental): Activa IM-Nail
  Interventions: Device: Activa IM-Nail

INTERVENTIONS:
Device: Activa IM-Nail — PLGA bioabsorbable intramedullary nail

SUMMARY:
Background

Pediatric diaphyseal forearm fractures are common and one of the most frequent reasons for orthopedic care. Fractures in need of surgery are often treated with metal Elastic Stable Intramedullary Nails (ESIN). Nail removal after 6-12 months is generally advocated. Surgical hardware removal has few complications; however, it is a substantial burden on the child, the family and healthcare economy. Bioabsorbable Intramedullary Nails (BIN) have been developed for the same indications as metal ESIN. The use of bioabsorbable implants would deem hardware removal unnecessary and relieve the child of further surgery and reduce healthcare costs.

Methods

The investigators aim to recruit all children in the catchment area of Herlev and Gentofte University Hospital (Copenhagen, Denmark) with acute unstable diaphyseal forearm fractures. Participants will be operated with BIN and followed consecutively for 2 years with interim analysis of data after 6 months. The investigators will report radiological healing using the Radiographic Union Score (RUS) 3 months after surgery together with any adverse events during follow-up.

Discussion

This study will provide important preliminary data and asses the feasibility of using the bioabsorbable Activa IM-Nail™ in pediatric diaphyseal forearm fractures. This study is a pilot study for initiating an RCT comparing BIN to metal ESIN hypothesizing that BIN is not an inferior treatment.

ELIGIBILITY:
Inclusion Criteria:

* Acute traumatic diaphyseal forearm fracture of the radius, ulna or both
* Fractures need to be complete (not unicortical or green stick)
* Displaced more than 50% of bone width or angulated more than 10° in any plane or irreducible or unstable after reduction

Exclusion Criteria:

We exclude patients

* with fractures that are well managed conservatively (undisplaced or minimally displaced)
* with previous ipsilateral forearm fracture
* with fractures unsuited for intramedullary nailing (e.g. multifragmentary, metaphyseal or epiphyseal)
* with fractures with ipsilateral wrist or elbow involvement (e.g. Monteggia or Galeazzi variants)
* unable to participate in follow-up
* with existing bone pathology (e.g. tumor, osteogenesis imperfecta, degenerative disease)
* in whom internal fixation is otherwise contraindicated (e.g. active or potential infection)

Ages: 2 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30 (Estimated)
Dates: Start 2021-05-25 (Actual); Primary Completion 2023-08-31 (Estimated); Study Completion 2025-05-25 (Estimated)

PRIMARY OUTCOMES:
Radiographic Union Score (RUS) | 3 months
  RUS is a score derived from assessing AP and lateral radiographs. Each bone cortex (anterior, posterior, medial and lateral) is assigned a score of 1 to 3. A cortex with a visible fracture line and no callus is given a score of 1, a cortex with callus but a visible fracture line is scored as 2 and a cortex with bridging callus and no visible fracture line is scored as 3. Scores are added to give a minimum score of 4 (definitely not healed) and a maximum of 12 (definitely healed). 12 is best.

SECONDARY OUTCOMES:
Faces Pain Scale - Revised (FPS-R) | 3 months
  To measure the outcome of pain in children below 8 years of age. Pain evaluated by the child selecting 1 of 6 faces that represents their feeling of pain. Faces are scored 0, 2, 4, 6, 8 or 10. Scale 0-10 with 2 point increments. 0 = no pain, 10= very much pain. 0 is best.
Bilateral elbow and forearm range of motion | 3 months
  Measured in degrees by goniometer
Visual Analogue Scale (VAS) | 3 months
  Pain evaluated by the child putting a mark on a 10 cm long line. Most left=no pain, most right=worst possible pain. Distance from most left to the child's mark is measured with a ruler. 1 mm = 1 point. Value is given with 1 decimal, e.g. 64 mm = 6,4 points.
  Scale 0.0-10.0. With 0 = no pain, 10= worst possible pain. 0 is best.

CONTACTS AND LOCATIONS:
Overall Officials: Morten J Andersen, MD, Principal Investigator
Locations (1):
- Herlev and Gentofte University Hospital, Herlev, Capital Region, Denmark

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-05-24): https://cdn.clinicaltrials.gov/large-docs/12/NCT04941612/Prot_SAP_000.pdf